CLINICAL TRIAL: NCT02017132
Title: The Effect of Pomegranate Extract on Anthropometric, Physiological and Biochemical Parameters in Human Volunteers: an 8 Week Parallel, Double Blinded, Placebo Controlled, Randomised Trial.
Brief Title: Effect of Pomegranate Extract Intake on Body Composition and Blood Pressure.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queen Margaret University (Other)
Collaborators: PomeGreat (Unknown)
Responsible Party: Principal Investigator, Angela Stockton, Ph.D. Researcher, Queen Margaret University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: POM-02Extr
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Obesity; Diabetes; Cardiovascular Disease
Keywords: Pomegranate; Blood pressure; Body composition; Weight-loss; Fat mass; Polyphenols; Quality of Life
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Cardiovascular Diseases; Weight Loss | interventions — pomegranate fruit rind

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pomegranate extract (Active Comparator): 1.1g pomegranate extract capsule administered daily to each participant for 8 weeks
  Interventions: Dietary Supplement: Pomegranate extract
- Placebo capsule (Placebo Comparator): 1.1g placebo capsule taken daily by each participant for 8 weeks

INTERVENTIONS:
Dietary Supplement: Pomegranate extract
  Other Names: Pomegreat PurePlus
  Arms: Pomegranate extract

SUMMARY:
Pomegranate has gained widespread popularity since the health effects of the whole fruit, as well as its juices and extracts, have been studied in relation to a variety of chronic conditions such as hypertension, diabetes, obesity, cancer and cardiovascular disease.

The fruit consists of peel, seeds and berries or arils. The peel is rich in minerals and compounds such as polyphenols, but is not an edible part of the plant. In order to harness the benefits of all parts of the fruit, the whole fruit can be crushed and powdered and then easily consumed as pomegranate extract capsules.

Pomegranate has been shown to be effective at reducing cardiovascular disease risk factors, particularly with respect to decreasing blood pressure and increasing insulin sensitivity. Dietary polyphenols may also suppress body fat growth. Recently, positive effects on fat reduction have been shown using pomegranate and its extracts. In animal models it has been shown for both extract and leaf that there were significant decrease in food consumption and body weight, inhibiting the development of obesity. In the few human studies, there appeared to be a trend towards a reduction in waist circumference and fat mass, plus a halt in body weight increase, for both juice and seed oil.

This parallel, double blinded, randomised, placebo controlled trial aims to confirm previous results concerning the effect of whole pomegranate fruit on biochemical and physiological markers using a new pomegranate extract and to conduct original work to explore its effect on body weight, measurements and fat mass. Any similar interventions have not been double blinded or used pomegranate in extract form. Changes in physiological and biochemical markers will also be investigated.

The study hypothesis is that pomegranate extract will reduce BMI and body weight, fat mass, body measurements and blood pressure.

DETAILED DESCRIPTION:
This is a parallel, double blinded, placebo controlled, randomised trial. It will be conducted over an 8 week intervention phase, plus a pre-intervention registration and preparation period. Participants will be randomly assigned to either the pomegranate extract or placebo groups. One capsule of Pomegranate or placebo will be taken after the same time daily meal with water for 8 weeks.

Participants will be asked to visit the clinical lab three times. The first visit will be for baseline measurements and a 24 hour urine sample before the intervention begins; the second in week 4 for measurements only and the final visit in week 8 for measurements and the last urine collection. Blood pressure and anthropometric measurements will be taken at each visit. Urine will only be collected pre and post intervention.

The health related Quality of Life Questionnaire (Rand 36) will be administered at both the initial and final visits. This series of questions covers eight spheres of health and has been proven to be scientifically robust having been used in over 200 health related scientific trials.

Three day diet diaries will be used for recording energy intake and to determine any fluctuations in dietary intake over the study period. These will be completed by participants in the pre-intervention week and then at week 4 of the intervention. Participants complete 2 diet diaries in total.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with a BMI within the range of 18-34.9 kg/m².

Exclusion Criteria:

* Taking medications for heart, liver or kidney disease, or diabetes;
* recent weight loss within 2 months preceding the study;
* pregnancy;
* lactation;
* allergies to pomegranate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Changes in measurements of body mass indicators | Week 0, 4, 8
  These indicators are:
  Body weight; height; BMI; waist, hip and mid-upper arm circumference; fat and fat free mass.

SECONDARY OUTCOMES:
Changes in blood pressure | Week 0, 4, 8
  Systolic and diastolic blood pressure are taken when volunteers are supine

OTHER OUTCOMES:
Changes in Quality of life | Week 0, 8
  Administered through the Rand 36 questionnaire
Changes in urinary polyphenol and FRAP levels | Week 0, 8
  Measured using the 24hr urine collection
Change in urinary cortisol-to-cortisone ratio | Week 0, 8
  Determined via the 24hr urine collection

CONTACTS AND LOCATIONS:
Overall Officials: Angela EV Stockton, MSc, Principal Investigator — Queen Margaret University
Locations (1):
- Queen Margaret University, Musselburgh, Edinburgh, United Kingdom